CLINICAL TRIAL: NCT05503043
Title: Effects of Intravenous Lidocaine on Serum miRNA-135a and Its Downstream Proteins Rock2 and Add1 in Elderly Patients Undergoing Non-cardiac Surgery Under General Anesthesia.
Brief Title: Effect of Intravenous Lidocaine on Serum miRNA-135a in Patients Undergoing Non-cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Li-Zhao
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Organ Protection
Keywords: lidocaine; postoperative cognitive dysfunction; miRNA-135a; Rock2; Add1
MeSH Terms: conditions — Postoperative Cognitive Complications; Hereditary Sensory and Autonomic Neuropathies | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the first hour, 1.5 mg/kg for the second hour, 0.7 mg/kg until the end of the surgery.
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Normal saline administered as a bolus and an infusion with identical volume and rate changes as the treatment group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the frst hour, 1.5 mg/kg for the second hour, 0.7 mg/kg until the end of the surgery.
  Arms: Lidocaine
Drug: Normal saline — Patients are received equal volumes of saline intravenously until the end of the surgery
  Arms: Normal saline

SUMMARY:
The purpose of this study is to investigate the effects of intravenous lidocaine on serum miRNA-135a and its downstream proteins Rock2 and Add1 in elderly patients undergoing non-cardiac under general anesthesia.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a major complication following surgeries and anesthesia, especially in elderly individuals. Lidocaine, an inexpensive, widely available, and relatively safe compound, is a local anesthetic that readily crosses the blood-brain barrier. Intravenous lidocaine can reduce the incidence of POCD. However, the mechanism is still unclear.

Rock2 and Add1, which are regulated by miRNA-135a, play a key role in learning, memory, and cognition.

The objective of this study is to investigate the efficacy of intravenous lidocaine on the incidence of early POCD, and the levels of Rock2, Add1, and miRNA-135a in elderly patients undergoing non-cardiac under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective non-cardiac surgery under general anesthesia
* ASA physical status II-III
* Aged ≥65 years

Exclusion Criteria:

* Serious heart, lung, liver and kidney diseases
* Central nervous system injury
* Mental illness and drug dependence
* On regular use of analgesic/sedative/antidepressant
* Unable to cooperate
* Allergy to lidocaine
* MMSE < 23 points

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline miRNA-135A at the end of surgery immediately and 1, 3days after surgery | at preoperation, at the end of surgery immediately, 1day and 3day after surgery
  Venous blood was extracted, and the serum miRNA-135a level of patients were detected by PCR and ELISA before surgery, at the end of surgery, 1day and 3day after surgery
Changes from Baseline Rock2 at the end of surgery immediately and 1, 3days after surgery | at preoperation, at the end of surgery immediately, 1day and 3day after surgery
  Venous blood was extracted, and the serum Rock2 level of patients were detected by PCR and ELISA before surgery, at the end of surgery, 1day and 3day after surgery
Changes from Baseline Add1 at the end of surgery immediately and 1, 3days after surgery | at preoperation, at the end of surgery immediately, 1day and 3day after surgery
  Venous blood was extracted, and the serum Add1 level of patients were detected by PCR and ELISA before surgery, at the end of surgery, 1day and 3day after surgery

SECONDARY OUTCOMES:
Changes from Baseline mini-mental state examination (MMSE) at the end of surgery immediately and 1, 3days after surgery | at preoperation,1day and 3day after surgery
  MMSE was performed

OTHER OUTCOMES:
Postoperative cognitive dysfunction (POCD) | at preoperation,1day and 3day after surgery
  the incidence of POCD

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhao, Principal Investigator — General Hospital of Ningxia Medical University

IPD SHARING:
Plan to Share IPD: Undecided